CLINICAL TRIAL: NCT07083401
Title: An Open-label, Randomized, Fed, Single-dose, 2-sequence, 2-period Crossover Study to Evaluate the Pharmacokinetics and Safety Between Single Oral Administration of "BR3006" and Co-administration of "BR3006A", "BR3006B" and "BR3006C" in Healthy Adult Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety Between "BR3006" and Co-administration of "BR3006A", "BR3006B", and "BR3006C" in Healthy Adult Volunteers (Fed)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-DPMC-CT-105
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Diabete Mellitus
Keywords: Dapagliflozin; Pioglitazone; Metformin HCl
MeSH Terms: conditions — Diabetes Mellitus | interventions — dapagliflozin; Pioglitazone; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (R1+R2+R3 / T) (Experimental): R1+R2+R3: BR3006A, BR3006B, and BR3006C; T:
  BR3006
  Interventions: Drug: Dapagliflozin 10 mg/Pioglitazone 30 mg/Metformin HCl 1000 mg; Drug: Dapagliflozin 10 mg; Drug: Pioglitazone 30 mg; Drug: Metformin HCl 1000 mg
- Sequence B (T / R1+R2+R3) (Experimental): T: BR3006; R1+R2+R3: BR3006A, BR3006B, and BR3006C
  Interventions: Drug: Dapagliflozin 10 mg/Pioglitazone 30 mg/Metformin HCl 1000 mg; Drug: Dapagliflozin 10 mg; Drug: Pioglitazone 30 mg; Drug: Metformin HCl 1000 mg

INTERVENTIONS:
Drug: Dapagliflozin 10 mg/Pioglitazone 30 mg/Metformin HCl 1000 mg — Orally administered once per day
  Other Names: BR3006
Drug: Dapagliflozin 10 mg — Orally administered once per day
  Other Names: BR3006A
Drug: Pioglitazone 30 mg — Orally administered once per day
  Other Names: BR3006B
Drug: Metformin HCl 1000 mg — Orally administered once per day
  Other Names: BR3006C

SUMMARY:
This was an open-label, randomized, fed, single-dose, 2-sequence, 2- period crossover study to evaluate the pharmacokinetics and safety between single oral administration of "BR3006" and co-administration of "BR3006A", "BR3006B," and "BR3006C" in healthy adult volunteers.

DETAILED DESCRIPTION:
A total of 40 healthy volunteers will be enrolled to evaluate the pharmacokinetics and safety profiles of the study drug (one combination tablet of dapagliflozin 10 mg/pioglitazone 30 mg/metformin HCl 1000 mg) and the comparator (co-administration of dapagliflozin 10 mg, pioglitazone 30 mg, and metformin HCl 1000 mg, one tablet each, respectively) while fed.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged over 19 at the time of consent
* Those who are eligible to participate in the clinical trial at the discretion of the principal investigator (or a subinvestigator) through laboratory tests such as hematology tests, blood chemistry tests, serology tests, urine tests, and electrocardiogram (ECG) tests that were planned/performed with specification to the investigational product.
* Those who provided written consent after receiving sufficient explanations and fully understood the objective and details of this clinical trial, the characteristics of the investigational product, and the expected adverse events.

Exclusion Criteria:

* Those who have administered investigational products within 6 months from the first dose administration date in another clinical trial (including bioequivalent studies) (The end of study date is based on the last dose administration date.)
* Those who have undergone gastrointestinal surgeries or have gastrointestinal diseases (except appendectomy or hernia surgery) that may affect the absorption of the investigational products
* Female subjects who are pregnant, suspected of pregnancy, or nursing

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-05 (Actual); Primary Completion 2026-07-05 (Estimated); Study Completion 2026-07-05 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic variable - AUCt | [Time Frame: From Day 1, 0 hour (pre-dose) to Day 3 after dose administration]
  Area under the drug concentration-time curve over the time interval of "BR3006"
Pharmacokinetic variable - Cmax | [Time Frame: From Day 1, 0 hour (pre-dose) to Day 3 after dose administration]
  Maximum plasma concentration of "BR3006"

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus Yangji Hospital, Seoul, Gwanak-gu, South Korea

IPD SHARING:
Plan to Share IPD: No